CLINICAL TRIAL: NCT00205933
Title: Behavioral Processes Underlying Reward Processing in Depression
Status: Completed | Type: Observational
Sponsor: Affective Neuroscience Laboratory (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Diego Pizzagalli, Principal Investigator, Harvard University
Other Study IDs: 2003-P-000994
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-11

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Depression; Bipolar Disorder; Reward Processing
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this project is to use behavioral techniques to investigate emotional processing in subjects with major depression and healthy comparison subjects.

DETAILED DESCRIPTION:
A promising strategy for parsing the heterogeneity of Major Depressive Disorder is to identify phenotypes characterized by reliable functional abnormalities. Anhedonia, the lack of reactivity to pleasurable stimuli, is considered a trait marker for depression. Using an objective behavioral task this project aims to investigate hedonic capacity in subjects meeting a DSM-IV diagnosis of Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

Depressed participants:

* Right-handed
* DSM-IV diagnosis of MDD
* Score of at least 17 on the 21-item HAM-D scale
* Absence of any psychotropic medications for at least 2 weeks (6 months for dopaminergic drugs (including methylphenidate), 6 weeks for fluoxetine, and 4 weeks for neuroleptics and benzodiazepines because of longer half-lives.)
* No current or past history of MDD with psychotic features
* Absence of any other Axis I or Axis II diagnosis (Including bipolar disorder and current or lifetime history of alcohol or substance abuse or dependence.) Particularly, subjects with a history of alcoholism and substance abuse will be excluded, since dopaminergic alterations have been reported in these conditions. Exclusion of patients with comorbid Axis I or Axis II diagnoses will be necessary as evidence exists of alteration in dopamine receptor density in detached personality and social phobia. The alteration of dopamine in the brain may in turn alter behavior.
* Absence of significant medical conditions
* Absence of ECT in the previous 6 months
* Ability to provide informed consent/authorization

Bipolar participants:

* Both genders and all ethnic origins
* Age between 18 and 64
* Right-handed
* DSM-IV diagnosis of Bipolar Disorder I or II
* Score of at least 17 on the 21-item Hamilton Depression Rating Scale (HAM-D)
* Absence of any psychotropic medications for at least 2 weeks (6 months for dopaminergic drugs (including methylphenidate), 6 weeks for fluoxetine, and 4 weeks for neuroleptics and benzodiazepines because of longer half-lives.)
* No current or past history of MDD with psychotic features
* Absence of any other Axis I or Axis II diagnosis (Including current or lifetime history of alcohol or substance abuse or dependence.) Particularly, subjects with a history of alcoholism and substance abuse will be excluded.
* Absence of significant medical conditions
* Absence of ECT in the previous 6 months
* Ability to provide informed consent/authorization

Control Participants:

* Right-handed
* Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse), as assessed by the SCID
* Absence of any medications for at least 2 weeks
* Informed consent/authorization

Exclusion Criteria:

* Left-handed/ambidextrous
* Evidence of neurological illness
* Current alcohol or substance abuse
* Serious suicide or homicide risk

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control participants, Participants with MDD, Participants with Bipolar Disorder
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2004-04; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Pizzagalli, PhD, Principal Investigator — Harvard University
Locations (2):
- United States (2):
  - The Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts
  - Affective Neuroscience Laboratory, Department of Psychology, Harvard University, Cambridge, Massachusetts